CLINICAL TRIAL: NCT02066181
Title: A Phase III, Double Blind, Randomized, Placebo-Controlled Trial of Sorafenib in Desmoid Tumors or Aggressive Fibromatosis (DT/DF)
Brief Title: Sorafenib Tosylate in Treating Patients With Desmoid Tumors or Aggressive Fibromatosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2014-00264; NCI-2014-00264 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA091105_A04PAMDREVW01; A091105; A091105 (Other: Alliance for Clinical Trials in Oncology); A091105 (Other: CTEP); R01FD005105 (FDA); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Desmoid Fibromatosis
MeSH Terms: conditions — Desmoid Tumors | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (sorafenib tosylate) (Experimental): Patients receive sorafenib tosylate PO QD on days 1-28.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Sorafenib Tosylate
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-28. Patients may crossover to Arm I upon disease progression.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Optional ancillary studies
  Other Names: Quality of Life Assessment
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
  Arms: Arm I (sorafenib tosylate)

SUMMARY:
This randomized phase III trial compares the effects, good and/or bad, of sorafenib tosylate in treating patients with desmoid tumors or aggressive fibromatosis. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the proteins needed for cell growth. [Funding Source - FDA OOPD]

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival (PFS) rates of patients with desmoid tumors (DT)/deep fibromatosis (DF) who receive either sorafenib (sorafenib tosylate) or placebo using a double-blinded randomized phase III study.

SECONDARY OBJECTIVES:

I. To assess toxicity. II. To assess time to surgical intervention. III. To assess tumor response rates and survival.

TERTIARY OBJECTIVES:

I. To evaluate changes in magnetic resonance imaging (MRI) Tesla (T)2 to predict (or correlate) with a biological effect such as tumor growth (by Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1), and pain palliation. (Correlative companion study) II. The mechanism of action of sorafenib in DT/DF remains unknown. In patients consenting to undergo the paired tumor biopsies (A091105-ST1), treatment induced changes will be quantified by histology, gene expression profiling, proteomic changes and selected interrogation of key pathways by western blot and reverse transcription-polymerase chain reaction (RT-PCR). (Correlative companion study) III. To collect archival tissue, baseline (tumor, blood) and day 8 (tumor, blood) specimens for basic science research (A091105-ST1). (Correlative companion study) IV. To assess patient-reported adverse events and quality of life (QOL) as measured by the Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) and the single-item overall Linear Analogue Self-Assessment (LASA) (A091105-HO1). (Correlative companion study) V. To assess pain palliation measured by the "worst pain" item of the Brief Pain Inventory Short Form (A091105-HO1). (Correlative companion study)

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive sorafenib tosylate orally (PO) once daily (QD) on days 1-28.

ARM II: Patients receive placebo PO QD on days 1-28. Patients may crossover to Arm I upon disease progression.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up annually for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have confirmation of DT/DF by local pathologist prior to registration
* Patients may have been treated with locoregional therapies such as major surgery, radiation, radiofrequency ablation, or cryosurgery provided this has been completed at least 4 weeks prior to registration and recovered from therapy related toxicity to less than CTCAE grade 2
* Patients may have been treated with cytotoxic, biologic (antibody), immune or experimental therapy, tyrosine kinase inhibitors, hormone inhibitors or nonsteroidal anti-inflammatory drugs (NSAIDs) provided this has been completed at least 4 weeks prior to registration (6 weeks for mitomycin and nitrosoureas) and recovered from any therapy related toxicity to less than CTCAE grade 2
* Patients with prior or current treatment of sorafenib are excluded
* No concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel); low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted; please note that drugs that strongly induce or inhibit cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) or are associated with a risk of torsades are not allowed; chronic concomitant treatment of CYP3A4 inducers is not allowed (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St. John's wort); as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product; the following drugs are strong inhibitors of CYP3A4 and are not allowed during the treatment with sorafenib:

  * Boceprevir
  * Indinavir
  * Nelfinavir
  * Lopinavir/ritonavir
  * Saquinavir
  * Telaprevir
  * Ritonavir
  * Clarithromycin
  * Conivaptan
  * Itraconazole
  * Ketoconazole
  * Mibefradil
  * Nefazodone
  * Posaconazole
  * Voriconazole
  * Telithromycin

    * Drugs with possible or conditional risk of torsades should be used with caution knowing that sorafenib could prolong the QT interval
* Chronic daily NSAID use as treatment for controlling desmoid tumors is not allowed, and should be stopped >= 3 days prior to registration; NSAIDS are allowed when used for desmoid tumor-related pain or for symptoms that are unrelated to desmoid disease (eg. headache, arthritis)
* Patients must have measurable disease
* Patients have to meet one of the following criteria to be eligible:

  * Disease determined unresectable or entailing unacceptably morbid surgery based on 1 or more of the following characteristics:

    * Multifocal disease
    * Disease in which there is involvement or inadequate plane from: neurovascular bundle, bone, skin, or viscera
    * Large size in relationship to location OR multi-compartment involvement
  * Progression by radiographic imaging (10% increase in size by RECIST v1.1 within 6 months of registration)
  * Patients with symptomatic disease which meets the following criteria Brief Pain Inventory (BPI) score greater than or equal to 3 AND one of the following:

    * Inability to control pain with NSAIDs and considering addition of narcotics OR
    * > 30% increase in current use of narcotics OR
    * Addition of a new opioid narcotic
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients who are pregnant or nursing are not eligible
* No patients with a history of cardiac disease: congestive heart failure > class II New York Heart Association (NYHA); active coronary artery disease (CAD) (myocardial infarction or unstable angina within 6 months prior to study entry)
* No patients with inadequately controlled hypertension (defined as a blood pressure of >= 150 mmHg systolic and/or >= 90 mmHg diastolic), or any prior history of hypertensive crisis or hypertensive encephalopathy
* No patients with clinically significant gastrointestinal (GI) bleeding or bleeding diathesis within 30 days prior to registration
* Absolute neutrophil count >= 1,500/mm^3
* Hemoglobin >= 8 g/dl
* Platelets >= 75,000/mm^3
* Total bilirubin =< 1.5 x upper limits of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST])/serum glutamate pyruvate transaminase (SGPT) (aspartate aminotransferase [ALT]) =< 1.5 x ULN
* Calculated creatinine clearance >= 50 mL/min using the Cockcroft-Gault equation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-03-21 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mrinal M Gounder, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (150):
- United States (149):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Reid Health, Richmond, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center - 68th Street Place, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Sovah Health Martinsville, Martinsville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mazza GL, Petersen MM, Ginos B, Langlais BT, Heon N, Gounder MM, Mahoney MR, Zoroufy AJ, Schwartz GK, Rogak LJ, Thanarajasingam G, Basch E, Dueck AC. Missing data strategies for the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) in Alliance A091105 and COMET-2. Qual Life Res. 2022 Apr;31(4):1069-1080. doi: 10.1007/s11136-021-02968-1. Epub 2021 Aug 21. PMID 34420143
- [Derived] Basch E, Becker C, Rogak LJ, Schrag D, Reeve BB, Spears P, Smith ML, Gounder MM, Mahoney MR, Schwartz GK, Bennett AV, Mendoza TR, Cleeland CS, Sloan JA, Bruner DW, Schwab G, Atkinson TM, Thanarajasingam G, Bertagnolli MM, Dueck AC. Composite grading algorithm for the National Cancer Institute's Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Clin Trials. 2021 Feb;18(1):104-114. doi: 10.1177/1740774520975120. Epub 2020 Dec 1. PMID 33258687
- [Derived] Gounder MM, Mahoney MR, Van Tine BA, Ravi V, Attia S, Deshpande HA, Gupta AA, Milhem MM, Conry RM, Movva S, Pishvaian MJ, Riedel RF, Sabagh T, Tap WD, Horvat N, Basch E, Schwartz LH, Maki RG, Agaram NP, Lefkowitz RA, Mazaheri Y, Yamashita R, Wright JJ, Dueck AC, Schwartz GK. Sorafenib for Advanced and Refractory Desmoid Tumors. N Engl J Med. 2018 Dec 20;379(25):2417-2428. doi: 10.1056/NEJMoa1805052. PMID 30575484
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Sorafenib Tosylate): Patients receive sorafenib tosylate PO QD on days 1-28, 400 mg/day
Period: Overall Study
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Placebo)
Started | 50 | 37
Crossed Over | 0 | 28
Completed | 49 | 36
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Placebo) | Total
Number analyzed (Participants) | 50 | 37 | 87
Age, Continuous [Median (Full Range); unit: years] | 37 [18 to 72] | 37 [21 to 67] | 37 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 26 | 60
  Male | 16 | 11 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 41 | 29 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival(PFS) Rate
Description: PFS is defined as the time from randomization to the first occurrence of progression or death due to any cause. If no event exists, the PFS will be censored at the last disease assessment. Data following cross over will be analyzed and summarized separately from the data from the main course of treatment for these patients in an exploratory and hypothesis generating manner. Intention to treat principles will be used. Patient disease status was evaluated using RECSIT v1.1. Patients ending treatment for symptomatic deterioration without radiographic evidence of PD, were classified as having PD. Otherwise, patients not yet showing disease progression were classified as having no progression at the most recent disease assessment and in the following cases: crossing over to receive sorafenib, date of first non-protocol directed anti-cancer therapy, lost to follow-up, withdrawal of consent, and changing imaging methods from that which was used at study entry.
Time Frame: Time from randomization to the first occurrence of progression or death due to any cause, assessed up to 3 years
Population: All patients that received treatment and were assessed for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Placebo)
Number analyzed (Participants) | 49 | 35
Participants
  Progressed or Died | 7 | 22
  Alive and Progression Free | 42 | 13
Statistical Analysis 1: Comparison: Arm I (Sorafenib Tosylate) vs Arm II (Placebo); Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 11.3, 95% CI 1-sided [lower limit 5.7]

2. Secondary Outcome: Incidence of Adverse Events, Using the Patient Reported Outcomes-Common Terminology Criteria in Adverse Events Version 4.0
Description: INCLUDED IN THE ADVERSE EVENTS PORTION OF THE RESULTS SECTION. Frequency tables, summary statistics, and categorical analysis will be used to compare the distributions of toxicity for patients treated with sorafenib tosylate vs placebo. Data for patients who have crossed over or having received surgical or radiotherapy intervention will be summarized independently from their primary course of study treatment in an exploratory and hypothesis generating manner.
Time Frame: Up to 3 years
Population: Per protocol, crossover patients are excluded/censored from secondary analysis and endpoints.
Measure: Count of Participants; unit: Participants
Groups:
- Crossover Patients: After progression from Arm II(Placebo), patients receive sorafenib tosylate PO QD on days 1-28. These patients are per protocol, excluded/censored from secondary analysis and endpoints.
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Placebo) | Crossover Patients
Number analyzed (Participants) | 49 | 36 | 0
Participants | 49 | 36 | 0

3. Secondary Outcome: Time to Surgical Intervention During Treatment
Description: A log rank test will be used to compare the distributions of time to surgical intervention between the two arms using a 2-sided test and alpha=0.05 level of significance. Kaplan-Meier methodology will be used to estimate various time points and 95% confidence intervals will be calculated for these estimates. Surgery will be classified by outcome (eg, complete-macroscopic, complete-microscopic, or partial), type, location (eg, limb), thereafter analyzed by categorical analysis and descriptive statistics. Non-parametric methods will be used, as appropriate. Too few patients had surgery during treatment to perform analysis.
Time Frame: Time between randomization to the patient undergoing therapeutic surgical resection for this disease, assessed up to 3 years
Population: Only the number of patients is presented due to the Protected Health Information as to the time to surgery for each of these individual patients. Crossover patients are per protocol, excluded/censored from secondary analysis and endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Placebo) | Crossover Patients
Number analyzed (Participants) | 49 | 36 | 0
Participants
  Had surgery during treatment | 1 | 1 | 0
  Didn't have surgery during treatment | 48 | 35 | 0

4. Secondary Outcome: Overall Survival
Description: Kaplan-Meier methodology and log rank tests will be used to compare overall survival between the groups at various time points (eg, 1 year rate, 2 year rate, etc) and 95% confidence intervals will be calculated for these estimates. Data following crossover will be analyzed and summarized separately from the main course of treatment for these patients in an exploratory and hypothesis generating manner.
Time Frame: Time between the date of randomization to until death, assessed up to 3 years
Population: All patients that started treatment and were assessed for survival. Crossover patients were excluded/censored from secondary analysis and endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Placebo) | Crossover Patients
Number analyzed (Participants) | 49 | 35 | 0
Participants
  Deaths | 1 | 0 | 0
  Alive | 48 | 35 | 0

5. Secondary Outcome: Best Objective Status Between the Two Treatment Arms According to Response Evaluation Criteria in Solid Tumors Version 1.1
Description: Compared between the two treatment arms and using the Cochran-Mantel-Haenszel test. Complete Response (CR): All of the following must be true: a. Disappearance of all target lesions. b. Each target lymph node must have reduction in short axis to <1.0 cm. Partial Response (PR): At least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the BSD. Patients on Arm II (placebo) who crossover are censored for Best Objective Status at the time of crossover.
Time Frame: Up to 3 years
Population: All patients that started treatment and were assessed for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Placebo)
Number analyzed (Participants) | 49 | 35
Participants
  CR | 1 | 0
  PR | 15 | 7
  Stable Diseaes or Progression | 33 | 28

6. Secondary Outcome: Duration of Response
Description: Kaplan Meier methodology will be used to estimate the distribution of duration of response and the log-rank test will be used to test for a difference in duration of response between the two arms. Patients on Arm II (placebo) who crossover are censored for Duration of Response at the time of crossover.
Time Frame: Time between first tumor response and progression, assessed up to 3 years
Population: All patients that started treatment and were assessed for response.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Placebo)
Number analyzed (Participants) | 49 | 35
Months | 14.7 [8.7 to 18.6] | 11.0 [4.8 to 12.8]

7. Other Pre Specified Outcome: Percent Change in Tumor Size by Response Evaluation Criteria in Solid Tumors Version 1.1 (Correlative Companion Study-Imaging Study)
Description: Best response (ordinal variable) and percent T2 signal change (continuous) will be correlated by Spearman?s rho.
Time Frame: Baseline up to 3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Percent Changes in MRI T2 Signal (Correlative Companion Study-Imaging Study)
Description: Percent T2 signal change (continuous) will be correlated by Spearman?s rho. The percent changes in MRI T2 signal from Week 8 to subsequent imaging will be compared between groups with > 30% pain palliation using t-test or a nonparametric alternative (e.g., Wilcoxon rank-sum test).
Time Frame: Baseline up to 3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Time to Pain Progression Measured by the ?Worst Pain? Item of the Brief Pain Inventory Short Form (Correlative Companion Study- A091105-H01 QOL Study)
Description: Defined as a >= 30% increase compared with baseline in the worst pain intensity score (BPI-SF ?worst pain? item) or either a >= 30% increase in the average daily use of any type of opioid narcotic or the addition of a new opioid narcotic compared with baseline. Estimated for each arm using Kaplan-Meier estimates and will be compared between arms using a log- rank test. Descriptive statistics will include means, standard deviations, medians, and ranges for each continuous or ordinal scale/subscale/item by group at each time point.
Time Frame: Date of randomization to the earliest date that pain progression is observed, assessed up to 12 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Time to Pain Palliation Measured by the ?Worst Pain? Item of the Brief Pain Inventory Short Form (Correlative Companion Study-A091105-H01 QOL Study)
Description: Defined at each time point as >= 30% decrease from baseline in the worst pain intensity score (BPI-SF ?worst pain? item), with neither a concomitant >= 30% increase in average daily use of any opioid narcotic, nor addition of any new opioid narcotic, relative to baseline. Estimated for each arm using Kaplan-Meier estimates and will be compared between arms using a log- rank test. Descriptive statistics will include means, standard deviations, medians, and ranges for each continuous or ordinal scale/subscale/item by group at each time point.
Time Frame: Date of randomization to the earliest date that confirmed pain palliation is observed, assessed up to 12 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Duration of Pain Palliation Measured by the ?Worst Pain? Item of the Brief Pain Inventory Short Form (Correlative Companion Study- A091105-H01 QOL Study)
Description: Defined for all patients who experience confirmed pain palliation. Descriptive statistics will include means, standard deviations, medians, and ranges for each continuous or ordinal scale/subscale/item by group at each time point. Descriptive graphical techniques will include mean plots by group for each continuous or ordinal scale/subscale/item. Relative frequencies of responses for each ordinal item will also be generated at each time point by group.
Time Frame: Time from the earliest date that confirmed pain palliation is observed to the earliest date that pain progression is observed, assessed up to 12 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Rate of Pain Palliation Measured by the ?Worst Pain? Item of the Brief Pain Inventory Short Form (Correlative Companion Study-A091105-H01 QOL Study)
Description: Rate of pain palliation at week 8 confirmed as week 12 will be compared between arms using a two-sided alpha=0.05 chi-squared tests at the time of the final analysis. Descriptive statistics will include means, standard deviations, medians, and ranges for each continuous or ordinal scale/subscale/item by group at each time point. Descriptive graphical techniques will include mean plots by group for each continuous or ordinal scale/subscale/item. Relative frequencies of responses for each ordinal item will also be generated at each time point by group.
Time Frame: Baseline up to 12 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Cadherin-associated Protein, Beta 1 (CTNNB1) Genotype (Correlative Companion Study-A091105-ST1 Study)
Description: Associations among the possible predictors of response to sorafenib and CTNNBI mutations will be examined using Fisher?s exact test, Kruskal-Wallis test, or Spearman?s correlation coefficient as appropriate. Strata will be compared by using the log-rank test. Multivariate models will be constructed by introducing all variables aforementioned simultaneously into the model and then eliminating variables using the backward selection method. P values will be two-tailed and considered significant at alpha 0.05.
Time Frame: Up to 3 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: False Discovery Rate (Correlative Companion Study- A091105-ST1 Study)
Description: Permutation testing of the same selection will be performed 1000 times and the sample group labels switched around in each permutation. A two-sided t-test will be used to identify differentially expressed genes on log transformed data and those with a twofold change. False discovery rate will be assessed by permutation testing (n = 1000) of the sample group labels. Enrichment will be assessed by one-sided Fisher?s exact test with estimated false discovery rate.
Time Frame: Up to day 8
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Treatment-specific Gene Expression Signature (Correlative Companion Study- A091105-ST1 Study)
Description: The analysis will identify over- and under-expressed genes in pre-treatment and day 8 biopsies as compared to all control samples.
Time Frame: Up to day 8
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Changes in Immunohistochemistry Score of Vascular Endothelial Growth Factor (Correlative Companion Study- A091105-ST1 Study)
Description: Compared by paired t-test. Quantitative changes will be correlated with disease status at 1 year by Fishers exact test.
Time Frame: Baseline up to day 8
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Changes in Immunohistochemistry Score of Platelet-derived Growth Factor Receptor (Correlative Companion Study- A091105-ST1 Study)
Description: Compared by paired t-test. Quantitative changes will be correlated with disease status at 1 year by Fishers exact test.
Time Frame: Baseline up to day 8
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Changes in Immunohistochemistry Score of Beta-catenin Cytoplasm/Nuclear Ratio (Correlative Companion Study- A091105-ST1 Study)
Description: Compared by paired t-test. Quantitative changes will be correlated with disease status at 1 year by Fishers exact test.
Time Frame: Baseline up to day 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 years
Groups:
- Crossover Group: Upon disease progression, patients treated with placebo will be allowed to crossover to the open label sorafenib arm.
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Placebo) | Crossover Group
All-Cause Mortality (participants affected / at risk) | 1/49 | 0/36 | 0/28
Serious Adverse Events (participants affected / at risk) | 11/49 | 6/36 | 5/28
Other Adverse Events (participants affected / at risk) | 49/49 | 34/36 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Sorafenib Tosylate) (N=49) | Arm II (Placebo) (N=36) | Crossover Group (N=28)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (5) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (4) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (8) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Sorafenib Tosylate) (N=49) | Arm II (Placebo) (N=36) | Crossover Group (N=28)
Anemia (Blood and lymphatic system disorders) | 9 (27) | 4 (18) | 5 (18)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 2 (14)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (22) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (5) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (3) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 2 (6)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (3)
Hypothyroidism (Endocrine disorders) | 1 (4) | 0 (0) | 1 (2)
Blurred vision (Eye disorders) | 1 (6) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (2) | 0 (0) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 3 (18) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 16 (136) | 13 (144) | 16 (132)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (10) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (15) | 1 (5)
Constipation (Gastrointestinal disorders) | 11 (67) | 4 (12) | 2 (15)
Dental caries (Gastrointestinal disorders) | 2 (5) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 27 (254) | 12 (115) | 17 (172)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (25) | 2 (15)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (6)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 1 (4) | 2 (6)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (22) | 3 (7) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4)
Mucositis oral (Gastrointestinal disorders) | 11 (70) | 6 (31) | 8 (45)
Nausea (Gastrointestinal disorders) | 25 (196) | 15 (160) | 17 (133)
Oral dysesthesia (Gastrointestinal disorders) | 1 (40) | 0 (0) | 1 (33)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (38)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (42) | 8 (26) | 8 (22)
Chills (General disorders) | 1 (1) | 0 (0) | 4 (11)
Edema limbs (General disorders) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 36 (461) | 23 (206) | 21 (241)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 1 (5) | 1 (1) | 1 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (23) | 2 (5) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (5) | 3 (17) | 1 (10)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 1 (1) | 1 (2)
Nail infection (Infections and infestations) | 1 (8) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 30 (142) | 7 (29) | 10 (44)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 3 (4) | 0 (0) | 2 (8)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (18) | 3 (4) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (3) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (44) | 4 (25) | 4 (25)
Alkaline phosphatase increased (Investigations) | 3 (9) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 6 (11) | 3 (16) | 7 (37)
Blood bilirubin increased (Investigations) | 5 (63) | 4 (10) | 1 (5)
Cholesterol high (Investigations) | 1 (8) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 1 (2) | 0 (0) | 1 (3)
Hemoglobin increased (Investigations) | 2 (4) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 5 (29) | 4 (8) | 2 (20)
Lipase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 3 (10) | 2 (6)
Neutrophil count decreased (Investigations) | 5 (24) | 2 (6) | 4 (11)
Platelet count decreased (Investigations) | 8 (51) | 1 (1) | 3 (19)
Weight gain (Investigations) | 0 (0) | 1 (13) | 1 (11)
Weight loss (Investigations) | 2 (46) | 2 (14) | 4 (61)
White blood cell decreased (Investigations) | 3 (27) | 6 (38) | 5 (51)
Anorexia (Metabolism and nutrition disorders) | 15 (161) | 9 (60) | 9 (91)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (4) | 1 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (29) | 3 (5) | 3 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (8) | 1 (1) | 3 (6)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (7) | 1 (2) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 2 (4) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (6) | 2 (14) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (14) | 1 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (7) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (173) | 9 (46) | 14 (79)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (23) | 2 (19) | 1 (11)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (7) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (32) | 4 (14) | 4 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (206) | 12 (54) | 12 (79)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (19) | 2 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (9) | 3 (4) | 1 (7)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (10) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (10) | 2 (2) | 1 (12)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 7 (41) | 8 (58)
Memory impairment (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 4 (16) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (6)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (35) | 1 (2) | 2 (14)
Phantom pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (12)
Spasticity (Nervous system disorders) | 1 (7) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (9) | 1 (7) | 2 (9)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (3) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 1 (20) | 1 (11)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (9) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 2 (20) | 0 (0) | 1 (8)
Menorrhagia (Reproductive system and breast disorders) | 2 (7) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (13) | 0 (0) | 1 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0) | 1 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (8) | 1 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (2) | 1 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (172) | 4 (17) | 7 (82)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (61) | 0 (0) | 3 (10)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 35 (327) | 9 (36) | 19 (213)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (23)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (30) | 0 (0) | 4 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (75) | 0 (0) | 2 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (86) | 1 (3) | 6 (39)
Scalp pain (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (22) | 2 (9)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 7 (33) | 5 (22) | 2 (17)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 2 (57)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 1 (2)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 31 (412) | 14 (83) | 16 (229)
Lymphedema (Vascular disorders) | 1 (21) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT02066181/Prot_SAP_000.pdf